CLINICAL TRIAL: NCT03079934
Title: Vascular Healing After Implantation of Bioresorbable Vascular Scaffold in Different Clinical Settings and Follow-up Time Points
Brief Title: Vascular Healing After BVS-implantation
Status: Completed | Type: Observational
Sponsor: LMU Klinikum (Other)
Collaborators: Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK) (Other)
Responsible Party: Principal Investigator, Prof. Dr. Julinda Mehilli, Director, Interventional cardiology, LMU Klinikum
Other Study IDs: MucC002-14
Record Dates: First submitted 2016-03-11; First posted 2017-03-15 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Coronary Heart Disease
Keywords: Bioresorbable vascular scaffold; Optical coherence tomography; strut coverage; acute coronary syndrome
MeSH Terms: conditions — Coronary Disease; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Absorb-BVS: Bioresorbable vascular scaffold implantation
  Interventions: Device: Absorb-BVS

INTERVENTIONS:
Device: Absorb-BVS — BVS patients undergoing optical coherence tomography examination at follow-up
  Other Names: Absorb

SUMMARY:
Evaluation of coronary artery vessel wall healing at different time points in patients undergoing implantion of bioresorbable vascular scaffold by using intravascular imaging.

In addition long-term clinical follow-ups are planned for all patients treated with Absorb in the institution

DETAILED DESCRIPTION:
OCT-guided evalutation of the coronary vessel wall, endovascular healing and bioresorbable vascular scaffolds at different time points. These results will be analysed in terms of clinical presentation, gender and age.

ELIGIBILITY:
Inclusion Criteria:

* optical coherence tomography examination after BVS-implantation

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data of patients who undergo OCT examination at different time points after BVS implantation will be analysed.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-09-20 (Actual)

PRIMARY OUTCOMES:
the amount of tissue coverage per strut level analysis at OCT | 7 weeks
  according to study protocol

SECONDARY OUTCOMES:
amount of diameter stenosis per strut in OCT examination | 7 weeks
  according to study protocol
amount of diameter stenosis per strut in OCT examination | 24 months
  according to study protocol
healing score in OCT examination | 7 weeks
  according to study protocol
healing score in OCT examination | 24 months
  according to study protocol
proportion of malapposed and protruding struts per stent in OCT examination | 7 weeks
  according to study protocol
proportion of malapposed and protruding struts per stent in OCT examination | 24 months
  according to study protocol

CONTACTS AND LOCATIONS:
Overall Officials: Julinda Mehilli, MD, Study Chair — Munich University Clinic
Locations (1):
- Munich University Clinic, Munich, Bavarian, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Baquet M, Brenner C, Wenzler M, Eickhoff M, David J, Brunner S, Theiss H, Massberg S, Guagliumi G, Mehilli J. Impact of Clinical Presentation on Early Vascular Healing After Bioresorbable Vascular Scaffold Implantation. J Interv Cardiol. 2017 Feb;30(1):16-23. doi: 10.1111/joic.12359. Epub 2016 Nov 28. PMID 27896843